CLINICAL TRIAL: NCT01703052
Title: A Placebo-controlled Double-blind Single and Repeated Ascending Dose Study to Investigate the Safety and Tolerability of Inhaled CHF 6001 in Healthy Volunteers
Brief Title: Safety and Tolerability of Inhaled CHF 6001 in Healthy Volunteers (HV)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-1006-PR-0048
Record Dates: First submitted 2012-04-02; First posted 2012-10-10 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CHF 6001 SD or placebo (Experimental): Single administration of CHF 6001 dose levels 1 to 7 or placebo
  Interventions: Drug: CHF 6001 SD or placebo
- CHF 6001 MD or placebo (Experimental): Multiple administration of CHF 6001 dose levels 1 to 5 or placebo
  Interventions: Drug: CHF 6001 MD or placebo

INTERVENTIONS:
Drug: CHF 6001 SD or placebo — Dry Powder Inhaler
  Other Names: CHF 6001 DPI
  Arms: CHF 6001 SD or placebo
Drug: CHF 6001 MD or placebo — Dry Powder Inhaler
  Other Names: CHF 6001 DPI
  Arms: CHF 6001 MD or placebo

SUMMARY:
This study is designed to investigate the safety, tolerability and pharmacokinetics of inhaled CHF 6001 after single and multiple doses in healthy volunteers.

DETAILED DESCRIPTION:
The study will be conducted in a single centre and will consist of a single dose part and a multiple dose part.

Seven single doses of CHF 6001 will be administered according to an escalation, alternate cross over scheme. Five multiple doses of CHF 6001 will be administered for 7 days according to a sequential escalation scheme.

ELIGIBILITY:
Inclusion Criteria:

* Subject's written informed consent obtained prior to any study-related procedure
* Male healthy volunteers aged 18-55 years;
* Able to understand the study procedures, the risks involved and ability to be trained to use the devices correctly.
* Body Mass Index (BMI) between 18.0 and 28.0 kg/m2;
* Non- or ex-smokers who smoked < 5 pack years (pack-years = the number of cigarette packs per day times the number of years) and stopped smoking > 1 year;
* Results of laboratory tests within the normal ranges. Minor deviations are acceptable provided that they are not judged clinically significant by the investigator.
* A reliable method of contraception for the subjects and their partner.

Exclusion Criteria:

* Blood donation or blood loss less than 8 weeks before inhalation of the study medication;
* Positive HIV1 or HIV2 serology;
* Positive results from the Hepatitis serology which indicates acute or chronic Hepatitis B or Hepatitis C;
* History of substance abuse or drug abuse within 12 months prior to screening visit or with a positive urine drug screen at screening;
* Clinically relevant abnormal laboratory values suggesting an unknown disease and requiring further clinical investigation;
* Clinically significant and uncontrolled cardiac, hepatic, renal, gastrointestinal, endocrine, metabolic, neurologic, or psychiatric disorder that may interfere with successful completion of this protocol;
* Treatment within the previous 3 months with any drug known to have a well defined potential for hepatotoxicity (e.g. isoniazide, nimesulide, ketoconazole).
* Subjects who refuse to abstain from alcohol or caffeine containing foods or beverages or grapefruit containing foods or beverages from 48 hour prior to each intake of study medication until the end of confinement at the clinical centre.
* Heavy caffeine drinker (> 5 cups or glasses of caffeinated beverages e.g., coffee, tea, cola per day).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2011-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Adverse events, adverse drug reactions, serious adverse events. | After 7 days of treatment
  The number and percentage of subjects with adverse events, adverse drug reactions, serious adverse events
Vital signs | After 7 days of treatment
  Blood pressure and Heart rate
12-lead ECG | After 7 days of treatment
  Heart rate, RR, PR, QRS, QT, QTcB, QTcF
24h ECG Holter | After 7 days of treatment
  Number and percentages of subjects with arrhythmias ( e.g ventricular tachycardia, supra ventricular tachycardia,..)
FEV1 | After 7 days of treatment
Blood and urine Laboratory tests | After 7 days of treatment
Body weight | After 7 days of treatment

SECONDARY OUTCOMES:
Pharmacokinetics of CHF 6001 and its metabolite | After 7 days of treatment
  AUC; Cmax and tmax; t½

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Mair, MD, Principal Investigator — Quotient Clinical
Locations (1):
- Quotient Clinical, Nottingham, United Kingdom

REFERENCES:
- [Background] Ferrari A, Compagnoni A, Nandeuil A, Maison-Blanche P. Evaluation of the Effects of CHF6001, an Inhaled PDE4 Inhibitor, on Cardiac Repolarization and Cardiac Arrhythmias in Healthy Volunteers. J Cardiovasc Pharmacol. 2016 Jul;68(1):41-8. doi: 10.1097/FJC.0000000000000384. PMID 26945156
- [Background] Jolling K, Abelo A, Luyckx N, Nandeuil MA, Govoni M, Cella M, Lindauer A. Concentration-QT Modeling Following Inhalation of the Novel Inhaled Phosphodiesterase-4 Inhibitor CHF6001 in Healthy Volunteers Shows an Absence of QT Prolongation. CPT Pharmacometrics Syst Pharmacol. 2019 Jul;8(7):460-468. doi: 10.1002/psp4.12405. Epub 2019 May 11. PMID 31077576
- [Result] Mariotti F, Govoni M, Lucci G, Santoro D, Nandeuil MA. Safety, tolerability, and pharmacokinetics of single and repeat ascending doses of CHF6001, a novel inhaled phosphodiesterase-4 inhibitor: two randomized trials in healthy volunteers. Int J Chron Obstruct Pulmon Dis. 2018 Oct 18;13:3399-3410. doi: 10.2147/COPD.S174156. eCollection 2018. PMID 30425469